CLINICAL TRIAL: NCT02345850
Title: A Randomized, Multi-Center, Phase III Trial of Calcineurin Inhibitor-Free Interventions for Prevention of Graft-versus-Host Disease (BMT CTN 1301; Progress II)
Brief Title: Calcineurin Inhibitor-Free Interventions BMT CTN 1301 for Prevention of Graft-versus-Host Disease (BMT CTN 1301)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: Blood and Marrow Transplant Clinical Trials Network (Network); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BMT CTN 1301; U01HL069294 (NIH)
Record Dates: First submitted 2015-01-22; First posted 2015-01-26 (Estimated); Results first posted 2021-12-21 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Acute Leukemia; Myelodysplasia
Keywords: Acute Leukemia; Myelodysplasia; GVHD Prophylaxis; Chronic GVHD
MeSH Terms: conditions — Anemia, Refractory, with Excess of Blasts; Bronchiolitis Obliterans Syndrome | interventions — Tacrolimus; Methotrexate; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tacrolimus/Methotrexate Control Arm (Active Comparator): Unmanipulated bone marrow graft with Tacrolimus/Methotrexate GVHD prophylaxis. Tacrolimus will be maintained at therapeutic doses for a minimum of 90 days. Methotrexate will be dosed at 5-15mg/m^2 for a maximum of 4 doses post-transplant.
  Cyclosporine may be substituted for tacrolimus if the patient is intolerant of tacrolimus or per institutional practice.
  Interventions: Procedure: Unmanipulated Bone Marrow Graft with Tacrolimus/Methotrexate; Drug: Tacrolimus; Drug: Methotrexate
- CD34 Selection Arm (Experimental): Mobilized CD34-selected Peripheral Blood Stem Cell graft
  Following screening and enrollment, the donor of patients randomized to the CD34-selection arm will receive mobilization therapy with once daily Granulocyte Colony Stimulating Factor (G-CSF). Mobilization will begin on Day -5 prior to the patient's transplant date.
  Leukapheresis will be performed on a continuous flow cell separator according to institutional standards and will commence on the morning of the fifth day of G-CSF treatment. The anti-coagulant used for the procedure will be acid citrate dextrose (ACD).
  Decisions concerning the need for further product collection will be based on the known or projected enriched CD34+ cell content of the previously collected products.
  Interventions: Procedure: Mobilized CD34-selected Peripheral Blood Stem Cell graft
- Post Transplant Cyclophosphamide (Experimental): Unmanipulated Bone Marrow Graft with Cyclophosphamide
  Interventions: Procedure: Unmanipulated Bone Marrow Graft with Cyclophosphamide; Drug: Cyclophosphamide

INTERVENTIONS:
Procedure: Unmanipulated Bone Marrow Graft with Tacrolimus/Methotrexate — Unmanipulated BM grafts will be administered on Day 0 to all patients according to individual institutional guidelines after appropriate processing and quantification has been performed by the local laboratory. Stem cells are administered through an indwelling central venous catheter. If infusion occurs over two days, Day 0 is the first day the infusion is initiated.
  Arms: Tacrolimus/Methotrexate Control Arm
Procedure: Mobilized CD34-selected Peripheral Blood Stem Cell graft — Mobilized CD34-selected PBSC grafts will be administered on Day 0 to all patients according to individual institutional guidelines after appropriate processing and quantification has been performed by the local laboratory. Stem cells are administered through an indwelling central venous catheter. If infusion occurs over two days, Day 0 is the first day the infusion is initiated.
  Arms: CD34 Selection Arm
Procedure: Unmanipulated Bone Marrow Graft with Cyclophosphamide — Unmanipulated BM grafts will be administered on Day 0 to all patients according to individual institutional guidelines after appropriate processing and quantification has been performed by the local laboratory. Stem cells are administered through an indwelling central venous catheter. If infusion occurs over two days, Day 0 is the first day the infusion is initiated.
  Arms: Post Transplant Cyclophosphamide
Drug: Cyclophosphamide — Mesna will be given in divided doses IV 30 min pre- and at 3, 6, and 8 hours post-cyclophosphamide or administered per institutional standards. Mesna dose will be based on the cyclophosphamide dose being given. The total daily dose of Mesna is equal to 80% of the total daily dose of cyclophosphamide.
  Cyclophosphamide 50 mg/kg will be given on Day 3 post-transplant (between 60 and 72 hours after marrow infusion) and on Day 4 post-transplant (approximately 24 hours after Day 3 cyclophosphamide). Cyclophosphamide will be given as an IV infusion over 1-2 hours (depending on volume).
  Other Names: Cytoxan®
  Arms: Post Transplant Cyclophosphamide
Drug: Tacrolimus — Tacrolimus will be given orally or intravenously per institutional standards starting Day -3. The dose of tacrolimus may be rounded to the nearest 0.5 mg for oral formulations. Subsequent dosing will be based on blood levels, with a target of 5-15 ng/ml. If patients are on medications which alter the metabolism of tacrolimus (e.g. azoles), the initial starting dose and subsequent doses should be altered as per institutional practices. Tacrolimus taper can be initiated at a minimum of 90 days post HSCT if there is no evidence of active GVHD. The rate of tapering will be done according institutional practices but patients should be off tacrolimus by Day 180 post HSCT if there is no evidence of active GVHD.
  Other Names: Prograf®; FK506
  Arms: Tacrolimus/Methotrexate Control Arm
Drug: Methotrexate — Methotrexate will be administered at the doses of 15 mg/m^2 IV bolus on Day +1, and 10 mg/m^2 IV bolus on Days +3, +6 and +11 after hematopoietic stem cell infusion. The Day +1 dose of methotrexate should be given at least 24 hours after the hematopoietic stem cell infusion. Dose reduction of MTX due to worsening creatinine clearance after initiation of conditioning regimen, high serum levels or development of oral mucositis is allowed according to institutional practices. Leucovorin rescue is allowed according to institutional practices.
  Other Names: MTX
  Arms: Tacrolimus/Methotrexate Control Arm

SUMMARY:
The study is designed as a three arm randomized Phase III, multicenter trial comparing two calcineurin inhibitor (CNI)-free strategies for Graft-versus-Host Disease (GVHD) prophylaxis to standard tacrolimus and methotrexate (Tac/Mtx) in patients with hematologic malignancies undergoing myeloablative conditioning hematopoietic stem cell transplantation.

DETAILED DESCRIPTION:
Chronic Graft-versus-Host Disease (GVHD) is a complication that affects many hematopoietic stem cell transplant (HSCT) survivors; it occurs when the new cells from a transplant attack the recipient's body. The current standard GVHD prophylaxis regimen for patients with hematologic malignancies undergoing HSCT involves a combination of immunosuppressive agents given for the first 6 months after transplant. Often, patients develop GVHD and continue on these agents for much longer periods. The combination of calcineurin inhibitors (tacrolimus and cyclosporine A) with methotrexate (MTX) is the most common GVHD prophylaxis used worldwide in the context of myeloablative conditioning transplants. This regimen demonstrates better control of acute GVHD, but is less effective against chronic GVHD. Management of chronic GVHD remains a challenge and it has become a significant health problem in transplant survivors with more frequent use of mobilized peripheral blood stem cells. Additionally, several issues arise with the standard approach including various toxicity symptoms and side effects, increased risk of thrombotic microangiopathy due to CNI, no prevention of other infectious diseases, and no prevention for disease relapse.

This standard strategy of Tac/MTX will be used as a control in comparison to two other treatment plans both utilizing CNI-free methods: CD34 selected T-cell depletion in peripheral blood stem cell (PBSC) grafts, and infusion of bone marrow (BM) grafts followed by post-transplant Cyclophosphamide (PTCy). Study participants will be randomized to one of these three treatment arms.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged ≥ 1.0 year and < 66.0 years
2. Patients with acute leukemia in morphologic complete remission with or without hematologic recovery or with myelodysplasia (MDS) with no circulating blasts and with less than 5% blasts in the bone marrow. Patients with CMML must have a WBC count ≤ 10,000 cells/µL and < 5% blasts in the marrow. Patients with ≥ 5% blasts due to a regenerating marrow must contact the protocol chairs for review.
3. Planned myeloablative conditioning regimen
4. Patients must have a related or unrelated donor as follows:

   1. Related donor must be an 8/8 match for human leukocyte antigen (HLA)-A, -B, and -C at intermediate (or higher) resolution, and -DRB1 at high resolution using DNA-based typing. Pediatric related donors must weigh ≥ 25.0 kg., must have adequate peripheral venous catheter access for leukapheresis or must agree to placement of a central catheter, must be willing to (1) donate bone marrow and (2) receive G-CSF followed by donation of peripheral blood stem cells (product to be determined by randomization post enrollment) and must meet institutional criteria for donation.
   2. Unrelated donor must be an 8/8 match at HLA-A, -B, -C and -DRB1 at high resolution using DNA-based typing. Unrelated donor must be medically eligible to donate according to National Marrow Donor Program (NMDP) (or equivalent donor search organization) criteria. At time of enrollment, the donor should not have any known preferences or contraindications to donate bone marrow or peripheral blood stem cells. (Selection of unrelated donors is to be performed according to institutional practice. It is recommended that the time from collection to initiation of the cell processing be considered when prioritizing donors, as data shows better results for CD34 selection when cell processing begins within 36 hours of the end of collection)
5. Cardiac function: Ejection fraction at rest ≥ 45.0% or shortening fraction of ≥ 27.0% by echocardiogram or radionuclide scan (MUGA).
6. Estimated creatinine clearance (for patients > 12 years) greater than 50.0 mL/minute (using the Cockcroft-Gault formula and actual body weight); for pediatric patients (> 1 year to 12 years), Glomerular Filtration Rate (GFR) estimated by the updated Schwartz formula ≥ 90.0 mL/min/1.73 m^2. If the estimated creatinine clearance is < 90 mL/min/1.73 m^2, then renal function must be measured by 24-hour creatinine clearance or nuclear GFR, and must be > 70.0 mL/min/1.73 m^2.
7. Pulmonary function: Diffusing capacity of the lung for carbon monoxide (DLCO) ≥ 50% (adjusted for hemoglobin), and forced expiratory volume in one second (FEV1) or forced vital capacity (FVC) ≥ 50%; for children who are unable to perform for Pulmonary Function Tests (PFTs) due to age or developmental ability, there must be no evidence of dyspnea and no need for supplemental oxygen, as evidenced by O2 saturation ≥ 92% on room air.
8. Liver function: total bilirubin < 2x the upper limit of normal (unless elevated bilirubin is attributed to Gilbert's Syndrome) and alanine aminotransferase (ALT) / aspartate aminotransferase (AST) < 2.5x the upper limit of normal.
9. Signed informed consent.

Exclusion Criteria:

1. Prior autologous or allogeneic hematopoietic stem cell transplant
2. Karnofsky or Lansky Performance Score < 70%
3. Active central nervous system (CNS) involvement by malignant cells
4. Patients with uncontrolled bacterial, viral or fungal infections (currently taking medication and with progression or no clinical improvement) at time of enrollment
5. Presence of fluid collection (ascites, pleural or pericardial effusion) that interferes with methotrexate clearance or makes methotrexate use contraindicated
6. Patients seropositive for HIV-1 or -2
7. Patients seropositive for Human T-Lymphotrophic Virus (HTLV)-I or -II
8. Patients with active Hepatitis B or C viral replication by polymerase chain reaction (PCR)
9. Documented allergy to iron dextran or murine proteins
10. Women who are pregnant (positive serum or urine βHCG) or breastfeeding
11. Females of childbearing potential (FCBP) or men who have sexual contact with FCBP unwilling to use 2 effective forms of birth control or abstinence for one year after transplantation
12. History of uncontrolled autoimmune disease or on active treatment
13. Patients with prior malignancies, except resected non-melanoma or treated cervical carcinoma in situ. Cancer treated with curative intent ≥ 5 years previously will be allowed. Cancer treated with curative intent < 5 years previously will not be allowed unless approved by the Protocol Officer or one of the Protocol Chairs.
14. Patient unable to comply with the treatment protocol including appropriate supportive care, follow-up and research tests
15. Planned post-transplant maintenance therapy except for FLT3 inhibitors or TKIs must be declared prior to randomization.
16. If it is known prior to enrollment that the hematopoietic stem cell product will need to be cryopreserved, the patient should not be enrolled.
17. German centers only: Treatment with any known non-marketed drug substance or experimental therapy within 5 terminal half lives or 4 weeks prior to enrollment, whichever is longer, or participation in any other interventional clinical study.

Ages: 1 Year to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 346 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2020-10-05 (Actual); Study Completion 2020-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Horowitz, MD, Study Director — Center for International Blood and Marrow Transplant Research
Locations (28):
- United States (28):
  - City of Hope National Medical Center, Duarte, California
  - Stanford Hospital and Clinics, Stanford, California
  - University of Florida College of Medicine, Gainesville, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Blood & Marrow Transplant Program at Northside Hospital, Atlanta, Georgia
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Hospital, Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Johns Hopkins/SKCCC, Baltimore, Maryland
  - Dana Farber Cancer Institute/Brigham & Women's, Boston, Massachusetts
  - Dana Farber Cancer Institute/Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Washington University/Barnes Jewish Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Weill Cornell Medical Center/New York Presbyterian, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - University Hospitals of Cleveland/Case Western, Cleveland, Ohio
  - Ohio State/Arthur G. James Cancer Hospital, Columbus, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Virginia Commonwealth University/MCV Hospitals, Richmond, Virginia
  - University of Wisconsin Hospital & Clinics, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Results will be published in a manuscript and supporting information submitted to NIH BioLINCC (including data dictionaries, case report forms, data submission documentation, documentation for outcomes dataset, etc where indicated).
Supporting Information: Study Protocol, ICF
Time Frame: Within 6 months of official study closure at participating sites.
Access Criteria: Available to the public
URL: https://biolincc.nhlbi.nih.gov/home/

REFERENCES:
- [Derived] Luznik L, Pasquini MC, Logan B, Soiffer RJ, Wu J, Devine SM, Geller N, Giralt S, Heslop HE, Horowitz MM, Jones RJ, Litzow MR, Mendizabal A, Muffly L, Nemecek ER, O'Donnell L, O'Reilly RJ, Palencia R, Schetelig J, Shune L, Solomon SR, Vasu S, Ho VT, Perales MA. Randomized Phase III BMT CTN Trial of Calcineurin Inhibitor-Free Chronic Graft-Versus-Host Disease Interventions in Myeloablative Hematopoietic Cell Transplantation for Hematologic Malignancies. J Clin Oncol. 2022 Feb 1;40(4):356-368. doi: 10.1200/JCO.21.02293. Epub 2021 Dec 2. PMID 34855460
- [Derived] Del Pozo Martin Y. 47th Annual Meeting of the EBMT. Lancet Haematol. 2021 May;8(5):e317-e318. doi: 10.1016/S2352-3026(21)00104-6. Epub 2021 Mar 31. No abstract available. PMID 33811823

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to accrual on August 17, 2015. Thirty-two participating centers were activated for enrollment and two of those were closed earlier without any enrollment. The study closed accrual on June 4, 2018 with 346 participants enrolled from 26 centers. Among the randomized participants, 327 participants received a transplant. Within the 19 participants who did not receive a transplant, there were 10 withdrawals of consents, 5 deaths, and 4 lost to follow-ups.
Groups:
- CD34 Selected Graft: Mobilized CD34-selected Peripheral Blood Stem Cell graft
  Following screening and enrollment, the donor of patients randomized to the CD34-selection arm will receive mobilization therapy with once daily Granulocyte Colony Stimulating Factor (G-CSF). Mobilization will begin on Day -5 prior to the patient's transplant date.
  Leukapheresis will be performed on a continuous flow cell separator according to institutional standards and will commence on the morning of the fifth day of G-CSF treatment. The anti-coagulant used for the procedure will be acid citrate dextrose (ACD).
  Decisions concerning the need for further product collection will be based on the known or projected enriched CD34+ cell content of the previously collected products.
  Mobilized CD34-selected Peripheral Blood Stem Cell graft: Mobilized CD34-selected PBSC grafts will be administered on Day 0 to all patients according to individual institutional guidelines after appropriate processing and quantification has been performed by the local laboratory. Stem cells are administered through an indwelling central venous catheter. If infusion occurs over two days, Day 0 is the first day the infusion is initiated.
- Post-Transplant Cyclophosphamide: Unmanipulated Bone Marrow Graft with Cyclophosphamide
  Unmanipulated BM grafts will be administered on Day 0 to all patients according to individual institutional guidelines after appropriate processing and quantification has been performed by the local laboratory. Stem cells are administered through an indwelling central venous catheter. If infusion occurs over two days, Day 0 is the first day the infusion is initiated.
  Cyclophosphamide: Mesna will be given in divided doses IV 30 min pre- and at 3, 6, and 8 hours post-cyclophosphamide or administered per institutional standards. Mesna dose will be based on the cyclophosphamide dose being given. The total daily dose of Mesna is equal to 80% of the total daily dose of cyclophosphamide.
  Cyclophosphamide 50 mg/kg will be given on Day 3 post-transplant (between 60 and 72 hours after marrow infusion) and on Day 4 post-transplant (approximately 24 hours after Day 3 cyclophosphamide). Cyclophosphamide will be given as an IV infusion over 1-2 hours (depending on volume).
- Tacrolimus/Methotrexate Control: Unmanipulated bone marrow graft with Tacrolimus/Methotrexate (Tac/MTX) GVHD prophylaxis. Tac will be maintained at therapeutic doses for a minimum of 90 days. Cyclosporine may be substituted for Tac if the patient is intolerant of tacrolimus or per institutional practice. MTX will be dosed at 10-15mg/m^2 for a maximum of 4 doses post-transplant.
  Tac will be given orally or intravenously per institutional standards starting Day -3. The dose of Tac may be rounded to the nearest 0.5 mg for oral formulations. Subsequent dosing will be based on blood levels, with a target of 5-15 ng/ml. If patients are on medications which alter the metabolism of Tac (e.g. azoles), the initial starting dose and subsequent doses should be altered as per institutional practices. Tac taper can be initiated at a minimum of 90 days post HSCT if there is no evidence of active GVHD. The rate of tapering will be done according institutional practices but patients should be off tacrolimus by Day 180 post HSCT if there is no evidence of active GVHD.
  MTX will be administered at the doses of 15 mg/m^2 IV bolus on Day +1, and 10 mg/m^2 IV bolus on Days +3, +6 and +11 after hematopoietic stem cell infusion. The Day +1 dose of MTX should be given at least 24 hours after the hematopoietic stem cell infusion. Dose reduction of MTX due to worsening creatinine clearance after initiation of conditioning regimen, high serum levels or development of oral mucositis is allowed according to institutional practices.
Period: Overall Study
Arm/Group | CD34 Selected Graft | Post-Transplant Cyclophosphamide | Tacrolimus/Methotrexate Control
Started | 114 | 114 | 118
Completed | 101 | 106 | 112
Not Completed | 13 | 8 | 6
Not completed — Not transplanted | 10 | 5 | 4
Not completed — Lost to Follow-up | 2 | 3 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are summarized for all patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | CD34 Selected Graft | Post-Transplant Cyclophosphamide | Tacrolimus/Methotrexate Control | Total
Number analyzed (Participants) | 114 | 114 | 118 | 346
Age, Continuous [Median (Full Range); unit: years] | 51.2 [21.9 to 66.0] | 50.9 [19.9 to 65.6] | 51.3 [13.1 to 64.6] | 51.1 [13.1 to 66.0]
Age, Customized [Count of Participants; unit: Participants]
  1-18 | 0 | 0 | 2 | 2
  19-40 | 29 | 28 | 28 | 85
  41-60 | 63 | 69 | 76 | 208
  >60 | 22 | 17 | 12 | 51
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 43 | 54 | 149
  Male | 62 | 71 | 64 | 197
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 7 | 7 | 21
  Not Hispanic or Latino | 105 | 102 | 107 | 314
  Unknown or Not Reported | 2 | 5 | 4 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 4 | 2 | 3 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 3 | 4 | 9
  White | 106 | 101 | 104 | 311
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 8 | 7 | 17
Lansky/Karnofsky Performance Score [Count of Participants; unit: Participants] — KPS describes patient-perceived global quality of life and functioning on a scale of 0-100.
  100: No evidence of disease; 90: Normal activity. Minor signs or symptoms of disease; 80: Normal activity with effort. Some signs or symptoms of disease; 70: Cares for self. Unable to continue normal activity; 60: Needs occasional assistance, but cares for most personal needs; 50: Needs considerable assistance and medical care; 40: Disabled. Needs special care and assistance; 30: Severely disabled. Hospital admission indicated; 20: Very sick. Active supportive therapy needed; 10: Moribund; 0: Dead
  Participants
    90-100 | 63 | 72 | 61 | 196
    70-80 | 51 | 42 | 57 | 150
Primary Disease [Count of Participants; unit: Participants]
  Acute Lymphoblastic Leukemia (ALL) | 30 | 27 | 23 | 80
  Acute Myelogenous Leukemia (AML) | 63 | 74 | 75 | 212
  Myelodysplastic Syndrome (MDS) | 19 | 11 | 16 | 46
  Chronic Myelomonocytic Leukemia (CMML) | 1 | 1 | 1 | 3
  Acute Undifferentiated Leukemia | 1 | 0 | 1 | 2
  Biphenotypic Leukemia | 0 | 1 | 2 | 3
Disease Risk [Count of Participants; unit: Participants] — Disease risk data was collected by CIBMTR. For AML and ALL: High risk (not in remission): Never treated, PIF, Relapse; Non-high: CR1, CR2 and CR3+.
  For MDS (including CMML): High risk: High risk: RAEB, RAEB-T, RAEB-1, RAEB-2, CMML; non-high: RA, RARS, RCMD, RCMD/RS, MDS Unclassifiable, isolated 5q- syndrome.
  Participants
    Non-high | 67 | 67 | 71 | 205
    High | 36 | 39 | 40 | 115
    Missing/Unknown | 11 | 8 | 7 | 26
Disease Stage for AML and ALL [Count of Participants; unit: Participants] — 1st CR: meet all for >=4 weeks: no blast cells in the peripheral blood, < 5% blasts in the bone marrow, no blasts with Auer rods, normal maturation of all cellular components in the marrow, normal CBC and ANC of > 1000/µL; Platelets ≥ 100000/µL; No other signs or symptoms of disease.
  >=2nd CR: after CR, relapsed and achieved CR again. Final is CR. PIF: recipient treated but never achieved durable CR. Relapse: ≥ 5% blasts in the marrow; Extramedullary disease; Reappearance of cytogenetic abnormalities and/or molecular markers associated with the diagnosis at a level representing relapse. Population: Disease Stage is assessed in patients diagnosed of AML or ALL .
  Participants
    number analyzed (Participants) | 93 | 101 | 98 | 292
    1st complete remission | 65 | 67 | 75 | 207
    >= 2nd complete remission | 15 | 21 | 15 | 51
    Relapse | 2 | 1 | 1 | 4
    Primary induction failure (PIF)/Untreated | 2 | 5 | 3 | 10
    Missing | 9 | 7 | 4 | 20
Donor type [Count of Participants; unit: Participants]
  Related Donor | 43 | 43 | 45 | 131
  Unrelated Donor | 71 | 71 | 73 | 215
Cytogenetic [Count of Participants; unit: Participants] — For Adult acute myeloid leukemia (AML), Favorable: t(15:17), inv(16), del(16q), t(16:16), [t(8:21) without del(9q) or complex]; Intermediate: normal karyotype, +6, +8, -Y, del(12p), 11q23, t(9:11); Poor: complex karyotype, -5/del(5q), -7/del(7q), abn(3q, 9q, 11q, 21q, 17p), t(6:9), t(9:22). For Acute lymphocytic leukemia (ALL), Poor: Ph+/t(9:22), t(4:11), 11q23, MLL, hypodiploid, t(8:14), complex. For Myelodysplastic Syndrome (MDS): Favorable: normal karyotype, isolated del(5q), del(20q), or -Y; Poor: complex karyotype, 7 chromosome abnormalities; Intermediate: other abnormalities.
  Participants
    Normal | 5 | 2 | 4 | 11
    Favorable | 13 | 12 | 12 | 37
    Intermediate | 50 | 54 | 56 | 160
    Poor | 35 | 38 | 39 | 112
    Missing | 11 | 8 | 6 | 25
    Not tested | 0 | 0 | 1 | 1
HLA matching 8/8 [Count of Participants; unit: Participants] | 114 | 114 | 118 | 346
Time from diagnosis to transplantation [Median (Full Range); unit: months] | 5.6 [1.9 to 121.7] | 4.7 [1.6 to 231.3] | 5.0 [1.9 to 139.7] | 5.0 [1.6 to 231.3]
HCT-comorbidity index [Count of Participants; unit: Participants] — The HCT-CI was developed to identify comorbidities relevant to transplant and act as a tool for risk assessment and before allogeneic hematopoietic stem cell transplantation. Patients with no comorbidities are assigned a score of zero. Arrhythmia, cardiac, bowel, diabetes, cerebrovascular, psychological, mild chronic hepatitis, obesity, infection are assigned a score of 1. Rheumatoid arthritis, peptic ulcer, renal moderate/severe, pulmonary moderate, are assigned a score of 2. Solid tumor, heart valve disease, pulmonary sever, hepatic moderate/severe are assigned a score of 3. Population: HCT-Comorbidity Index Score is assessed in transplanted patients.
  Participants
    number analyzed (Participants) | 104 | 109 | 114 | 327
    0 | 38 | 41 | 44 | 123
    1-2 | 37 | 43 | 49 | 129
    3 or greater | 29 | 25 | 21 | 75
Pre-Transplant CMV status [Count of Participants; unit: Participants] — Population: Pre-Transplant CMV Status is assessed in transplanted patients.
  Participants
    number analyzed (Participants) | 104 | 109 | 114 | 327
    Positive | 45 | 54 | 57 | 156
    Negative | 59 | 55 | 57 | 171
Donor CMV Status [Count of Participants; unit: Participants] — Population: Donor CMV Status is assessed in transplanted patients.
  Participants
    number analyzed (Participants) | 104 | 109 | 114 | 327
    Negative | 73 | 55 | 71 | 199
    Positive | 31 | 53 | 43 | 127
    Unknown | 0 | 1 | 0 | 1
Stem cell source [Count of Participants; unit: Participants] — Population: Stem cell source is assessed in transplanted patients.
  Participants
    number analyzed (Participants) | 104 | 109 | 114 | 327
    Peripheral Blood | 98 | 11 | 12 | 121
    Bone Marrow | 6 | 98 | 102 | 206

OUTCOME MEASURES:

1. Primary Outcome: Chronic GVHD-free, Relapse-free Survival (CRFS) Probability
Description: The primary endpoint of the trial is Chronic GVHD/Relapse-Free Survival (CRFS), treated as a time to event variable. An event for this time to event outcome is defined as moderate to severe chronic GVHD, disease relapse, or death by any cause. Participant will be censored if lost to follow up prior to 2 years. Time is from randomization to the event of moderate to severe chronic GVHD, disease relapse, death, last follow up, or 2 years, whichever comes first. The primary analysis is performed using the intent-to-treat principle (ITT) so that all randomized patients are included in the analysis.
Time Frame: 2 years
Population: All randomized patients are analyzed for this endpoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CD34 Selected Graft | Post-Transplant Cyclophosphamide | Tacrolimus/Methotrexate Control
Number analyzed (Participants) | 114 | 114 | 118
percentage of participants
  1 year Post Randomization | 60.2 [50.3 to 68.7] | 60.3 [50.5 to 68.7] | 52.6 [43.1 to 61.3]
  2 years Post Randomization | 50.6 [40.8 to 59.6] | 48.1 [38.5 to 57.1] | 41.0 [32.0 to 49.9]
Statistical Analysis 1: Comparison: CD34 Selected Graft vs Tacrolimus/Methotrexate Control; The primary null hypothesis of the study is that there is no difference of the CRFS hazard ratio between CD34 select graft vs. Tac/MTX Control. The data in primary outcome table provides point estimates at specific time points (1 year and 2 years post randomization). The statistics in this session provides comparisons between different arms for the entire period of the study; Test type: Superiority; p = 0.2368, Log Rank — The primary pairwise comparisons are tested at a Bonferroni adjusted significance level of 0.05/3; Hazard Ratio (HR) = 0.805, 95% CI 2-sided [0.562 to 1.154]
Statistical Analysis 2: Comparison: Post-Transplant Cyclophosphamide vs Tacrolimus/Methotrexate Control; The primary null hypothesis of the study is that there is no difference of the CRFS hazard ratio between Post-Transplant Cyclophosphamide vs. Tac/MTX Control. The data in primary outcome table provides point estimates. The statistics in this session provides comparisons between different arms for the entire period of the study; Test type: Superiority; p = 0.4134, Log Rank — The primary pairwise comparisons are tested at a Bonferroni adjusted significance level of 0.05/3; Hazard Ratio (HR) = 0.864, 95% CI 2-sided [0.609 to 1.228]
Statistical Analysis 3: Comparison: CD34 Selected Graft vs Post-Transplant Cyclophosphamide; The primary null hypothesis of the study is that there is no difference of the CRFS hazard ratio between CD34 select graft vs. Post-Transplant Cyclophosphamide. The data in primary outcome table provides point estimates. The statistics in this session provides comparisons between different arms for the entire period of the study; Test type: Superiority; p = 0.7166, Log Rank — The primary pairwise comparisons are tested at a Bonferroni adjusted significance level of 0.05/3; Hazard Ratio (HR) = 0.933, 95% CI 2-sided [0.643 to 1.355]
Statistical Analysis 4: Comparison: CD34 Selected Graft vs Post-Transplant Cyclophosphamide vs Tacrolimus/Methotrexate Control; The null hypothesis is that there is no difference of the CRFS hazard ratio between treatment groups after adjustment for age, donor type, performance status, primary disease, and disease risk. The data in primary outcome table provides point estimates. The statistics in this session provides comparisons between different arms for the entire period of the study; Test type: Superiority; p = 0.386, Regression, Cox — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 5: Comparison: CD34 Selected Graft vs Post-Transplant Cyclophosphamide vs Tacrolimus/Methotrexate Control; Subgroup analyses are conducted for CRFS according to disease, disease risk and age. Interaction tests between treatment group and subgroup are conducted within a Cox proportional hazards regression model with treatment, subgroup, and a treatment*subgroup interaction term. The null hypothesis is that there is no Interaction between treatment group and disease risk (Low/Intermediate vs. High) for CRFS; Test type: Superiority; p = 0.461, Cox proportional hazards regression — A Bonferroni adjusted significance level of 0.05/3=0.0167 is used for each of three interaction tests to account for multiple testing
Statistical Analysis 6: Comparison: CD34 Selected Graft vs Post-Transplant Cyclophosphamide vs Tacrolimus/Methotrexate Control; Subgroup analyses are conducted for CRFS according to disease, disease risk and age. Interaction tests between treatment group and subgroup are conducted within a Cox proportional hazards regression model with treatment, subgroup, and a treatment*subgroup interaction term. The null hypothesis is that there is no Interaction between treatment group and Age (<=50 vs. >50) for CRFS; Test type: Superiority; p = 0.115, Cox proportional hazards regression — Cox proportional hazards regression
Statistical Analysis 7: Comparison: CD34 Selected Graft vs Post-Transplant Cyclophosphamide vs Tacrolimus/Methotrexate Control; Subgroup analyses are conducted for CRFS according to disease, disease risk and age. Interaction tests between treatment group and subgroup are conducted within a Cox proportional hazards regression model with treatment, subgroup, and a treatment*subgroup interaction term. The null hypothesis is that there is no Interaction between treatment group and Disease (AML vs. ALL vs. MDS) for CRFS; Test type: Superiority; p = 0.227, Cox proportional hazards regression — [p-value comment as in outcome 1, analysis 5]

2. Secondary Outcome: Percentage of Participants With Overall Survival (OS)
Description: OS is a key secondary endpoint, with explicit control of the type I error rate through a gatekeeper approach. Formal significance testing of OS between a CNI-free strategy and the control will be conducted if the corresponding CRFS comparison is significant. This OS comparison will be done using a Bonferroni adjusted significance level of 0.05/3 to account for three potential CNI-free comparisons to the control. Otherwise, survival analyses will be considered exploratory. Death from any cause is considered as event for this endpoint. Participant is censored if lost to follow up.
Time Frame: 2 Years
Population: The randomized or transplanted participants are included in the analyses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CD34 Selected Graft | Post-Transplant Cyclophosphamide | Tacrolimus/Methotrexate Control
Number analyzed (Participants) | 114 | 114 | 118
percentage of participants
  1 year post-randomization | 75.7 [66.4 to 82.8] | 84.6 [76.4 to 90.1] | 84.2 [76.1 to 89.7]
  2 year post-randomization | 60.1 [50.1 to 68.8] | 76.2 [67.1 to 83.1] | 76.1 [67.2 to 83.0]
  1 year post-transplantation: number analyzed (Participants) | 104 | 109 | 114
  1 year post-transplantation | 74.8 [65.2 to 82.1] | 83.4 [74.9 to 89.2] | 83.3 [75.0 to 89.0]
  2 year post-transplantation: number analyzed (Participants) | 104 | 109 | 114
  2 year post-transplantation | 61.6 [51.4 to 70.3] | 76.7 [67.5 to 83.6] | 74.2 [65.0 to 81.3]
Statistical Analysis 1: Comparison: CD34 Selected Graft vs Tacrolimus/Methotrexate Control; The null hypothesis is that there is no difference of the OS hazard ratio between CD34 select graft vs. Tac/MTX Control; Test type: Superiority; p = 0.0197, Log Rank — The OS pairwise comparisons are tested at a Bonferroni adjusted significance level of 0.05/3; Hazard Ratio (HR) = 1.744, 95% CI 2-sided [1.086 to 2.800]
Statistical Analysis 2: Comparison: Post-Transplant Cyclophosphamide vs Tacrolimus/Methotrexate Control; The null hypothesis is that there is no difference of the OS hazard ratio between Post-Transplant Cyclophosphamide vs. Tac/MTX Control; Test type: Superiority; p = 0.9525, Log Rank — The OS pairwise comparisons are tested at a Bonferroni adjusted significance level of 0.05/3; Hazard Ratio (HR) = 1.016, 95% CI 2-sided [0.599 to 1.724]
Statistical Analysis 3: Comparison: CD34 Selected Graft vs Post-Transplant Cyclophosphamide; The null hypothesis is that there is no difference of the OS hazard ratio between CD34 select graft vs. Post-Transplant Cyclophosphamide; Test type: Superiority; p = 0.0185, Log Rank — The OS pairwise comparisons are tested at a Bonferroni adjusted significance level of 0.05/3; Hazard Ratio (HR) = 1.774, 95% CI 2-sided [1.093 to 2.877]
Statistical Analysis 4: Comparison: CD34 Selected Graft vs Post-Transplant Cyclophosphamide vs Tacrolimus/Methotrexate Control; The null hypothesis is that there is no difference of the OS hazard ratio between treatment groups after adjustment for age, donor type, performance status, primary disease, and disease risk; Test type: Superiority; p = 0.026, Regression, Cox — Statistical significance was determined using a pre-specified threshold of 0.05

3. Secondary Outcome: Percentage of Participants With Relapse-free Survival
Description: The events for this endpoint RFS are death and relapse of the underlying malignancy. The analyses of this endpoint use the transplanted populations and time is from transplant to the event of disease relapse or death, or last follow up, whichever comes first.
Time Frame: 2 Years
Population: The analyses of this endpoint will use the transplanted population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CD34 Selected Graft | Post-Transplant Cyclophosphamide | Tacrolimus/Methotrexate Control
Number analyzed (Participants) | 104 | 109 | 114
percentage of participants
  1 year post-transplantation | 64.1 [54.0 to 72.5] | 78.8 [69.9 to 85.4] | 70.1 [60.8 to 77.6]
  2 years post-transplantation | 57.1 [46.9 to 66.0] | 70.3 [60.7 to 78.0] | 66.5 [56.9 to 74.3]
Statistical Analysis 1: Comparison: CD34 Selected Graft vs Post-Transplant Cyclophosphamide vs Tacrolimus/Methotrexate Control; The null hypothesis is that there is no difference of Relapse-Free Survival between the treatment groups; Test type: Superiority; p = 0.029, Log Rank — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 2: Comparison: CD34 Selected Graft vs Post-Transplant Cyclophosphamide vs Tacrolimus/Methotrexate Control; The null hypothesis is that there is no difference of the RFS hazard ratio between treatment groups after adjustment for age, donor type, performance status, primary disease, and disease risk; Test type: Superiority; p = 0.145, Regression, Cox — Statistical significance was determined using a pre-specified threshold of 0.05

4. Secondary Outcome: Percentage of Participants With Treatment-related Mortality
Description: The events for this endpoint TRM are deaths prior to relapse of the underlying malignancy. The analyses of this endpoint will use the transplanted populations, and time will be from transplant to the first of disease relapse, death, or last follow up. TRM are evaluated using the cumulative incidence function. Deaths without relapse are the events for this endpoint and relapse is a competing risk for this endpoint.
Time Frame: 2 Years
Population: The analyses of this endpoint will use the transplanted populations.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CD34 Selected Graft | Post-Transplant Cyclophosphamide | Tacrolimus/Methotrexate Control
Number analyzed (Participants) | 104 | 109 | 114
percentage of participants
  1 year post-transplantation | 16.5 [10.1 to 24.3] | 12.0 [6.7 to 18.9] | 7.0 [3.2 to 12.7]
  2 years post-transplantation | 21.5 [14.1 to 30.0] | 15.7 [9.6 to 23.2] | 7.9 [3.9 to 13.8]
Statistical Analysis 1: Comparison: CD34 Selected Graft vs Post-Transplant Cyclophosphamide vs Tacrolimus/Methotrexate Control; The null hypothesis is that there is no difference of Transplant-Related Mortality between the treatment groups; Test type: Superiority; p = 0.020, Gray's test for cumulative Incidence — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 2: Comparison: CD34 Selected Graft vs Post-Transplant Cyclophosphamide vs Tacrolimus/Methotrexate Control; The null hypothesis is that there is no difference of the TRM hazard ratio between treatment groups after adjustment for age, donor type, performance status, primary disease, and disease risk; Test type: Superiority; p = 0.040, Regression, Cox — Statistical significance was determined using a pre-specified threshold of 0.05

5. Secondary Outcome: Participants With Immunosuppression-free Survival
Description: Patients who are alive, relapse-free, and do not need ongoing immune suppression to control GVHD at one year post HSCT are considered successes for this endpoint. Immune suppression is defined as any systemic agents used to control or suppress GVHD.
Time Frame: 1 Year
Population: The analyses of this endpoint will use the transplanted populations. Two participant of CD34 Selected Graft arm and one participants of Post-Transplant Cyclophosphamide arm were lost to follow-up while alive and not relapsed, and they are considered as not evaluable for this endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | CD34 Selected Graft | Post-Transplant Cyclophosphamide | Tacrolimus/Methotrexate Control
Number analyzed (Participants) | 102 | 108 | 114
Participants | 59 | 73 | 66
Statistical Analysis 1: Comparison: CD34 Selected Graft vs Post-Transplant Cyclophosphamide vs Tacrolimus/Methotrexate Control; The null hypothesis is that there is no difference of immunosuppression-free survival at 1-year post-transplant between the treatment groups; Test type: Superiority; p = 0.2389, Chi-squared — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 2: Comparison: CD34 Selected Graft vs Post-Transplant Cyclophosphamide vs Tacrolimus/Methotrexate Control; The null hypothesis is that there is no agreement between CRFS and immunosuppression-free survival at 1-year post-transplant; Test type: Superiority; p < 0.0001, Cohen's Kappa

6. Secondary Outcome: Percentage of Participants With Disease Relapse
Description: Relapse is defined by either morphological evidence of acute leukemia or MDS consistent with pre-transplant features, or radiologic evidence of lymphoma, documented or not by biopsy. The event is defined as increase in size of prior sites of disease or evidence of new sites of disease, documented or not by biopsy. Relapse is adjudicated by ERC. Disease relapse is analyzed using cumulative incidence function with death as a competing risk. The analyses of this endpoint use the transplanted populations, and the time will be measured from transplant to the earliest of death, relapse/progression, or last follow up.
Time Frame: 2 Years
Population: The analyses of this endpoint use the transplanted populations.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CD34 Selected Graft | Post-Transplant Cyclophosphamide | Tacrolimus/Methotrexate Control
Number analyzed (Participants) | 104 | 109 | 114
percentage of participants
  1 year post transplantation | 19.4 [12.4 to 27.6] | 9.2 [4.7 to 15.6] | 22.9 [15.6 to 31.0]
  2 years post transplantation | 21.4 [14.0 to 29.8] | 13.9 [8.1 to 21.2] | 25.6 [17.9 to 33.9]
Statistical Analysis 1: Comparison: CD34 Selected Graft vs Post-Transplant Cyclophosphamide vs Tacrolimus/Methotrexate Control; The null hypothesis is that there is no difference of Disease Relapse between the treatment groups; Test type: Superiority; p = 0.076, Gray's test for cumulative Incidence — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 2: Comparison: CD34 Selected Graft vs Post-Transplant Cyclophosphamide vs Tacrolimus/Methotrexate Control; The null hypothesis is that there is no difference of the Disease Relapse hazard ratio between treatment groups after adjustment for age, donor type, performance status, primary disease, and disease risk; Test type: Superiority; p = 0.106, Regression, Cox — Statistical significance was determined using a pre-specified threshold of 0.05

7. Secondary Outcome: Percentage of Participants With Neutrophil Engraftment
Description: Neutrophil recovery is defined as achieving an absolute neutrophil count (ANC) ≥ 500/mm^3 for three consecutive measurements on three different days. The first of the three days will be designated the day of neutrophil recovery. The competing event is death without neutrophil recovery.
Time Frame: Day 28
Population: The analyses of the endpoint use the transplanted populations.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CD34 Selected Graft | Post-Transplant Cyclophosphamide | Tacrolimus/Methotrexate Control
Number analyzed (Participants) | 104 | 109 | 114
percentage of participants | 97.1 [90.5 to 99.1] | 91.7 [84.4 to 95.7] | 96.5 [90.3 to 98.8]
Statistical Analysis 1: Comparison: CD34 Selected Graft vs Post-Transplant Cyclophosphamide vs Tacrolimus/Methotrexate Control; The null hypothesis is that there is no difference of Neutrophil Engraftment post-transplantation between the treatment groups; Test type: Superiority; p = 0.0764, Gray's test for cumulative Incidence — Statistical significance was determined using a pre-specified threshold of 0.05

8. Secondary Outcome: Percentage of Participants With Platelet Recovery
Description: Platelet recovery is defined as the first day of a sustained platelet count >20,000/mm^3 with no platelet transfusion in the preceding seven days. The first day of sustained platelet count above this threshold will be designated the day of platelet engraftment. The competing event is death without platelet recovery.
Time Frame: Day 60
Population: The analyses of the endpoint use the transplanted populations. Three transplanted participants (one from the CD34 arm and two from the PTCy arm) are missing platelet data and are not included in the analyses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CD34 Selected Graft | Post-Transplant Cyclophosphamide | Tacrolimus/Methotrexate Control
Number analyzed (Participants) | 103 | 107 | 114
percentage of participants | 94.2 [86.9 to 97.5] | 91.6 [84.2 to 95.6] | 98.2 [93.4 to 99.9]
Statistical Analysis 1: Comparison: CD34 Selected Graft vs Post-Transplant Cyclophosphamide vs Tacrolimus/Methotrexate Control; The null hypothesis is that there is no difference of Platelet recovery post-transplantation between the treatment groups; Test type: Superiority; p = 0.0001, Gray's test for cumulative Incidence — Statistical significance was determined using a pre-specified threshold of 0.05

9. Secondary Outcome: Participants With Primary Graft Failure
Description: Primary graft failure is defined as no neutrophil recovery to > 500 cells/µL by Day 28 post HSCT.
Time Frame: Day 28
Population: The analyses of the endpoint use the transplanted populations.
Measure: Count of Participants; unit: Participants
Arm/Group | CD34 Selected Graft | Post-Transplant Cyclophosphamide | Tacrolimus/Methotrexate Control
Number analyzed (Participants) | 104 | 109 | 114
Participants | 3 | 9 | 4

10. Secondary Outcome: Percentage of Participants With Secondary Graft Failure
Description: Secondary graft failure will be assessed according to neutrophil count after initial hematologic recovery. Secondary graft failure is defined as initial neutrophil engraftment followed by subsequent decline in absolute neutrophil counts < 500 cells/µL, unresponsive to growth factor therapy, but cannot be explained by disease relapse or medications. Secondary graft failure will be analyzed using cumulative incidence function with death as a competing risk.
Time Frame: 2 Years
Population: The analyses of the endpoint use the transplanted populations.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CD34 Selected Graft | Post-Transplant Cyclophosphamide | Tacrolimus/Methotrexate Control
Number analyzed (Participants) | 104 | 109 | 114
percentage of participants | 2.9 [0.8 to 7.5] | 0 [0 to 0] | 0.9 [0.1 to 4.3]
Statistical Analysis 1: Comparison: CD34 Selected Graft vs Post-Transplant Cyclophosphamide vs Tacrolimus/Methotrexate Control; The null hypothesis is that there is no difference of Secondary graft failure post-transplantation between the treatment groups; Test type: Superiority; p = 0.1478, Gray's test for cumulative Incidence

11. Secondary Outcome: Percentage of Participants With Acute GVHD
Description: Cumulative incidences of grade II-IV and III-IV acute GVHD were determined. Death prior to acute GVHD is treated as the competing risk. Grading of acute GVHD was derived by consensus grading (Przepiorka 1995) per BMTCTN manual of procedures (MOP). The acute GVHD algorithm calculates the grade based on the organ (skin, GI and liver) stage and etiology/biopsy reported on the weekly GVHD form. Staging for skin: Stage 1. <25% rash; 2. 25-50%; 3. >50%; 4. generalized erythroderma with bullae. Staging for GI: Stage 1. Diarrhea>500ml/d or persistent nausea; 2. >1000ml/d; 3. >1500ml/d; 4. Large volume diarrhea and severe abdominal pain +- ileus. Staging for Liver: Stage 1. bilirubin 2-3mg/dl; 2. bilirubin 3-6 mg/dl; 3. bilirubin 6-15 mg/dl; 4. bilirubin>15mg/dl. Grade 4 is the worst outcome.
Time Frame: Day 100
Population: The analyses of the endpoint use the transplanted populations.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CD34 Selected Graft | Post-Transplant Cyclophosphamide | Tacrolimus/Methotrexate Control
Number analyzed (Participants) | 104 | 109 | 114
percentage of participants
  grade II-IV acute GVHD | 16.3 [9.9 to 24.1] | 37.6 [28.5 to 46.6] | 29.8 [21.7 to 38.4]
  grade III-IV acute GVHD | 2.9 [0.8 to 7.5] | 10.1 [5.3 to 16.6] | 3.5 [1.1 to 8.1]
Statistical Analysis 1: Comparison: CD34 Selected Graft vs Post-Transplant Cyclophosphamide vs Tacrolimus/Methotrexate Control; The null hypothesis is that there is no difference of grade II-IV acute GVHD post-transplantation between the treatment groups; Test type: Superiority; p = 0.0026, Gray's test for cumulative Incidence — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 2: Comparison: CD34 Selected Graft vs Post-Transplant Cyclophosphamide vs Tacrolimus/Methotrexate Control; The null hypothesis is that there is no difference of grade III-IV acute GVHD post-transplantation between the treatment groups; Test type: Superiority; p = 0.0369, Gray's test for cumulative Incidence — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 3: Comparison: CD34 Selected Graft vs Post-Transplant Cyclophosphamide vs Tacrolimus/Methotrexate Control; The null hypothesis is that there is no difference of the grade II-IV acute GVHD hazard ratio between treatment groups after adjustment for age, donor type, performance status, primary disease, and disease risk; Test type: Superiority; p = 0.002, Regression, Cox — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 4: Comparison: CD34 Selected Graft vs Post-Transplant Cyclophosphamide vs Tacrolimus/Methotrexate Control; The null hypothesis is that there is no difference of the grade III-IV acute GVHD hazard ratio between treatment groups after adjustment for age, donor type, performance status, primary disease, and disease risk; Test type: Superiority; p = 0.046, Regression, Cox — Statistical significance was determined using a pre-specified threshold of 0.05

12. Secondary Outcome: Participants With Maximum Acute GVHD
Description: Grading of acute GVHD was derived by consensus grading (Przepiorka 1995) per BMTCTN manual of procedures (MOP). The acute GVHD algorithm calculates the grade based on the organ (skin, GI and liver) stage and etiology/biopsy reported on the weekly GVHD form. Grade I aGVHD is defined as Skin stage of 1-2 and stage 0 for both GI and liver organs. Grade II aGVHD is stage 3 of skin, or stage 1 of GI, or stage 1 of liver. Grade III is stage 2-4 for GI, or stage 2-3 of liver. Grade IV is stage 4 of skin, or stage 4 of liver. Max acute GVHD by Day 100 was computed.
Time Frame: Day 100
Population: The analyses of the endpoint use the transplanted populations.
Measure: Count of Participants; unit: Participants
Arm/Group | CD34 Selected Graft | Post-Transplant Cyclophosphamide | Tacrolimus/Methotrexate Control
Number analyzed (Participants) | 104 | 109 | 114
Participants
  Grade 0, No aGVHD | 72 | 45 | 55
  Grade I | 15 | 23 | 25
  Grade II | 14 | 30 | 30
  Grade III | 3 | 9 | 4
  Grade IV | 0 | 2 | 0

13. Secondary Outcome: Percentage of Participants With Chronic GVHD
Description: The cumulative incidence of chronic GVHD will be determined. Death prior to acute GVHD is treated as the competing risk. Data will be collected directly from providers and chart review according to the recommendations of the NIH Consensus Criteria. Eight organs will be scored on a 0-3 scale to reflect degree of chronic GVHD involvement. Liver and pulmonary function test results and use of systemic therapy for treatment of chronic GVHD will also be recorded. This secondary endpoint of chronic GVHD will include mild, moderate and severe chronic GVHD based on NIH Consensus Criteria.
Time Frame: 2 Years
Population: The analyses of the endpoint use the transplanted populations.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CD34 Selected Graft | Post-Transplant Cyclophosphamide | Tacrolimus/Methotrexate Control
Number analyzed (Participants) | 104 | 109 | 114
percentage of participants
  1 year post-transplantation | 16.4 [9.8 to 24.5] | 33.0 [24.0 to 42.3] | 31.1 [22.5 to 40.1]
  2 years post-transplantation | 18.5 [11.5 to 26.8] | 37.0 [27.6 to 46.4] | 40.0 [30.5 to 49.3]
Statistical Analysis 1: Comparison: CD34 Selected Graft vs Post-Transplant Cyclophosphamide vs Tacrolimus/Methotrexate Control; The null hypothesis is that there is no difference of chronic GVHD post-transplantation between the treatment groups; Test type: Superiority; p = 0.0024, Gray's test for cumulative Incidence — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 2: Comparison: CD34 Selected Graft vs Post-Transplant Cyclophosphamide vs Tacrolimus/Methotrexate Control; The null hypothesis is that there is no difference of the chronic GVHD hazard ratio between treatment groups after adjustment for age, donor type, performance status, primary disease, and disease risk; Test type: Superiority; p = 0.005, Regression, Cox — Statistical significance was determined using a pre-specified threshold of 0.05

14. Secondary Outcome: Percentage of Participants With Chronic GVHD-free Survival
Description: The event for this endpoint includes moderate to severe chronic GVHD according to NIH consensus criteria global score, or death by any cause.
Time Frame: 2 Years
Population: The analyses of the endpoint use the transplanted populations.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CD34 Selected Graft | Post-Transplant Cyclophosphamide | Tacrolimus/Methotrexate Control
Number analyzed (Participants) | 104 | 109 | 114
percentage of participants
  1 year post-transplantation | 71.0 [61.4 to 78.6] | 67.4 [57.8 to 75.3] | 65.8 [56.3 to 73.7]
  2 years post-transplantation | 55.4 [45.3 to 64.3] | 54.2 [44.4 to 63.0] | 47.1 [37.7 to 56.0]
Statistical Analysis 1: Comparison: CD34 Selected Graft vs Post-Transplant Cyclophosphamide vs Tacrolimus/Methotrexate Control; The null hypothesis is that there is no difference of Chronic GVHD-free Survival post-transplantation between the treatment groups; Test type: Superiority; p = 0.229, Log Rank — Statistical significance was determined using a pre-specified threshold of 0.05

15. Secondary Outcome: Participants With Grade ≥ 3 Toxicity
Description: All grades ≥ 3 toxicities according to CTCAE, version 4 will be tabulated for each intervention arm. The number of unique patients is counted.
Time Frame: 2 Years
Population: The analyses of the endpoint use the transplanted populations.
Measure: Count of Participants; unit: Participants
Arm/Group | CD34 Selected Graft | Post-Transplant Cyclophosphamide | Tacrolimus/Methotrexate Control
Number analyzed (Participants) | 104 | 109 | 114
Participants
  Any Grade 3-5 Stem Cell Infusional Toxicities | 6 | 4 | 17
  Grades 3-5 Oral mucositis | 39 | 51 | 63
  Grades 3-5 Cystitis noninfective | 4 | 11 | 2
  Grades 3-5 Acute kidney injury | 12 | 13 | 15
  Grades 3-5 Chronic kidney disease | 4 | 4 | 3
  Grades 3-5 Hemorrhage | 12 | 9 | 4
  Grades 3-5 Hypotension | 19 | 15 | 11
  Grades 3-5 Hypertension | 20 | 21 | 30
  Grades 3-5 Cardiac arrhythmia | 9 | 6 | 8
  Grades 3-5 Left ventricular systolic dysfunction | 5 | 2 | 8
  Grades 3-5 Somnolence | 7 | 4 | 4
  Grades 3-5 Seizure | 6 | 0 | 2
  Grades 3-5 Thrombotic thrombocytopenic purpura | 1 | 2 | 4
  Grades 3-5 Capillary leak syndrome | 1 | 0 | 1
  Grades 3-5 Hypoxia | 32 | 22 | 14
  Grades 3-5 Dsypnea | 23 | 15 | 12
  Grades 3-4 ALT | 10 | 26 | 18
  Grades 3-4 AST | 11 | 27 | 19
  Grades 3-4 Bilirubin | 8 | 14 | 7
  Grades 3-4 Alkaline Phosphatase | 11 | 12 | 6
  Received dialysis | 5 | 2 | 6
  Abnormal liver function | 12 | 14 | 24
  SOS/VOD | 0 | 2 | 1
  IPS | 2 | 2 | 3
  Toxicities Within Day 100 | 68 | 82 | 81
  Toxicities Day 100 to 1 year | 26 | 33 | 41
  Toxicities 1 year to 2 years | 23 | 18 | 24
  Overall NCI CTCAE Grade 3-5 Toxicities | 80 | 88 | 100

16. Secondary Outcome: Participants Infected Post Transplant
Description: All grade 2 and grade 3 infections, as defined by the BMT CTN Technical MOP, occurring post transplantation will be reported. The incidence of definite and probable viral, fungal and bacterial infections will be tabulated for each intervention arm.
Time Frame: 2 Years
Population: The analyses of the endpoint use the transplanted populations.
Measure: Count of Participants; unit: Participants
Arm/Group | CD34 Selected Graft | Post-Transplant Cyclophosphamide | Tacrolimus/Methotrexate Control
Number analyzed (Participants) | 104 | 109 | 114
Participants
  Patients with Grades 2-3 infections | 72 | 66 | 50
  Patients with Grades 3 infections | 31 | 23 | 16
Statistical Analysis 1: Comparison: CD34 Selected Graft vs Post-Transplant Cyclophosphamide vs Tacrolimus/Methotrexate Control; The null hypothesis is that there is no difference of Grades II-III infection post-transplantation between the treatment groups; Test type: Superiority; p = 0.0006, Gray's test for cumulative Incidence — Superiority - Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 2: Comparison: CD34 Selected Graft vs Post-Transplant Cyclophosphamide vs Tacrolimus/Methotrexate Control; The null hypothesis is that there is no difference of Grades III infection post-transplantation between the treatment groups; Test type: Superiority; p = 0.0145, Gray's test for cumulative Incidence — Statistical significance was determined using a pre-specified threshold of 0.05

17. Secondary Outcome: Incidence of Infections
Description: as for outcome 16
Time Frame: 2 years
Population: The analyses of the endpoint use the transplanted populations.
Measure: Number; unit: number of Infection Events
Arm/Group | CD34 Selected Graft | Post-Transplant Cyclophosphamide | Tacrolimus/Methotrexate Control
Number analyzed (Participants) | 104 | 109 | 114
number of Infection Events | 157 | 161 | 123

18. Secondary Outcome: Health-Related Quality of Life (HQL) - Medical Outcomes Study Short Form 36 (SF36)
Description: HQL will be measured post-transplant using patient-reported survey SF36. The SF36 is a 36 item general assessment of health quality of life with eight components: Physical Functioning, Role Physical, Pain Index, General Health Perceptions, Vitality, Social Functioning, Role Emotional, Mental Health Index. Each domain is positively scored, indicating that higher scores are associated with positive outcome. The total score ranges from 0 to 100. This scale is being used in this protocol as a generic measure of quality of life. To facilitate comparison of results with published norms, the Physical Component Summary and Mental Component Summary are used as the outcome measures in summarizing the SF36 data. These summary scores are derived by multiplying the z-score for each scale by its respective physical or mental factor score coefficient and summing the products. Resulting scores are then transformed into Tscores (mean=50; standard deviation=10). The SF36 takes 6 minutes to complete.
Time Frame: Baseline, Day 100, Day 180, 1 year, 2 years
Population: The analyses of the endpoint use the transplanted populations.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CD34 Selected Graft | Post-Transplant Cyclophosphamide | Tacrolimus/Methotrexate Control
Number analyzed (Participants) | 104 | 109 | 114
score on a scale
  STANDARDIZED MENTAL COMPONENT SCALE at Baseline: number analyzed (Participants) | 86 | 75 | 68
  STANDARDIZED MENTAL COMPONENT SCALE at Baseline | 48 (1.0) | 46 (1.2) | 48 (1.1)
  STANDARDIZED MENTAL COMPONENT SCALE at Day 100: number analyzed (Participants) | 72 | 80 | 80
  STANDARDIZED MENTAL COMPONENT SCALE at Day 100 | 48 (1.0) | 48 (1.1) | 48 (1.0)
  STANDARDIZED MENTAL COMPONENT SCALE at Day 180: number analyzed (Participants) | 71 | 81 | 88
  STANDARDIZED MENTAL COMPONENT SCALE at Day 180 | 50 (1.1) | 50 (1.1) | 49 (0.9)
  STANDARDIZED MENTAL COMPONENT SCALE at 1 year: number analyzed (Participants) | 64 | 72 | 81
  STANDARDIZED MENTAL COMPONENT SCALE at 1 year | 50 (1.2) | 52 (1.1) | 49 (1.2)
  STANDARDIZED MENTAL COMPONENT SCALE at 2 years: number analyzed (Participants) | 48 | 55 | 66
  STANDARDIZED MENTAL COMPONENT SCALE at 2 years | 50 (1.5) | 50 (1.5) | 51 (1.1)
  STANDARDIZED PHYSICAL COMPONENT SCALE at Baseline: number analyzed (Participants) | 86 | 75 | 68
  STANDARDIZED PHYSICAL COMPONENT SCALE at Baseline | 42 (1.0) | 44 (1.0) | 41 (1.2)
  STANDARDIZED PHYSICAL COMPONENT SCALE at Day 100: number analyzed (Participants) | 72 | 80 | 80
  STANDARDIZED PHYSICAL COMPONENT SCALE at Day 100 | 40 (1.1) | 41 (1.1) | 40 (1.0)
  STANDARDIZED PHYSICAL COMPONENT SCALE at Day 180: number analyzed (Participants) | 71 | 81 | 88
  STANDARDIZED PHYSICAL COMPONENT SCALE at Day 180 | 43 (1.1) | 44 (1.2) | 44 (0.9)
  STANDARDIZED PHYSICAL COMPONENT SCALE at 1 year: number analyzed (Participants) | 64 | 72 | 81
  STANDARDIZED PHYSICAL COMPONENT SCALE at 1 year | 46 (1.2) | 47 (1.2) | 44 (1.1)
  STANDARDIZED PHYSICAL COMPONENT SCALE at 2 years: number analyzed (Participants) | 48 | 55 | 66
  STANDARDIZED PHYSICAL COMPONENT SCALE at 2 years | 46 (1.4) | 47 (1.2) | 47 (1.3)

19. Secondary Outcome: Health-Related Quality of Life (HQL) - Functional Assessment of Cancer Therapy - Bone Marrow Transplant (FACT-BMT)
Description: The FACT-BMT is a 37 item scale comprised of a general core questionnaire, the FACT-G with a possible range of 0-108 points, that evaluates the health-related quality of life (HQL) of patients receiving treatment for cancer, and a specific module, BMT Concerns, that addresses disease and treatment-related questions specific to bone marrow transplant. The FACT-G consists of four subscales developed and normed in cancer patients: Physical Well-being, Social/Family Well-being, Emotional Wellbeing, and Functional Well-being. Each subscale is positively scored, with higher scores indicating better functioning. The FACT-BMT Trial Outcome Index, comprised of the physical well-being scale, the functional well-being scale and the BMT specific items, will be used as the outcome measure in summarizing the FACT-BMT data. The FACT-BMT takes 6 minutes to complete. The final score for FACT-BMT ranges from 0 to 196. Higher scores for the scales and subscales indicate better quality of life.
Time Frame: Baseline, Day 100, Day 180, 1 year, 2 years
Population: The analyses of the endpoint use the transplanted populations.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CD34 Selected Graft | Post-Transplant Cyclophosphamide | Tacrolimus/Methotrexate Control
Number analyzed (Participants) | 104 | 109 | 114
score on a scale
  FACT-G Total at Baseline: number analyzed (Participants) | 86 | 79 | 70
  FACT-G Total at Baseline | 81 (1.6) | 79 (1.4) | 80 (1.9)
  FACT-G Total at Day 100: number analyzed (Participants) | 71 | 82 | 78
  FACT-G Total at Day 100 | 79 (1.7) | 80 (1.5) | 79 (1.6)
  FACT-G Total at Day 180: number analyzed (Participants) | 70 | 82 | 91
  FACT-G Total at Day 180 | 80 (1.9) | 83 (1.7) | 82 (1.6)
  FACT-G Total at 1 Year: number analyzed (Participants) | 61 | 74 | 84
  FACT-G Total at 1 Year | 84 (2.1) | 86 (2.0) | 84 (1.7)
  FACT-G Total at 2 Years: number analyzed (Participants) | 48 | 57 | 68
  FACT-G Total at 2 Years | 87 (2.5) | 86 (2.1) | 84 (2.1)
  FACT-BMT Trial Outcome Index at Baseline: number analyzed (Participants) | 86 | 78 | 70
  FACT-BMT Trial Outcome Index at Baseline | 67 (1.6) | 67 (1.3) | 65 (1.8)
  FACT-BMT Trial Outcome Index at Day 100: number analyzed (Participants) | 72 | 81 | 76
  FACT-BMT Trial Outcome Index at Day 100 | 63 (1.9) | 66 (1.5) | 63 (1.6)
  FACT-BMT Trial Outcome Index at Day 180: number analyzed (Participants) | 70 | 81 | 89
  FACT-BMT Trial Outcome Index at Day 180 | 67 (1.8) | 69 (1.8) | 67 (1.5)
  FACT-BMT Trial Outcome Index at 1 Year: number analyzed (Participants) | 61 | 73 | 84
  FACT-BMT Trial Outcome Index at 1 Year | 73 (1.9) | 72 (2.0) | 69 (1.7)
  FACT-BMT Trial Outcome Index at 2 Years: number analyzed (Participants) | 46 | 57 | 69
  FACT-BMT Trial Outcome Index at 2 Years | 73 (2.3) | 73 (2.1) | 71 (2.0)
  FACT-BMT Total at Baseline: number analyzed (Participants) | 86 | 77 | 70
  FACT-BMT Total at Baseline | 109 (2.1) | 108 (1.8) | 108 (2.4)
  FACT-BMT Total at Day 100: number analyzed (Participants) | 71 | 81 | 76
  FACT-BMT Total at Day 100 | 106 (2.4) | 108 (2.0) | 105 (2.2)
  FACT-BMT Total at Day 180: number analyzed (Participants) | 70 | 81 | 90
  FACT-BMT Total at Day 180 | 108 (2.5) | 112 (2.3) | 110 (2.1)
  FACT-BMT Total at 1 Year: number analyzed (Participants) | 61 | 73 | 84
  FACT-BMT Total at 1 Year | 114 (2.8) | 116 (2.6) | 113 (2.2)
  FACT-BMT Total at 2 Years: number analyzed (Participants) | 46 | 57 | 68
  FACT-BMT Total at 2 Years | 117 (3.4) | 115 (2.8) | 113 (2.7)

20. Secondary Outcome: Health-Related Quality of Life (HQL) - MDASI
Description: HQL will be measured post-transplant using patient-reported survey MD Anderson Symptom Inventory (MDASI). The MDASI is a 19 item instrument that captures 13 symptoms (0="not present" to 10="as bad as you can imagine") and 6 items measuring interference with life from 0 ("did not interfere") to 10 ("interfered completely"). MDASI Tool questions are negatively scored - higher levels indicate more severe symptoms and levels of interference. Codelist for each question is from 0 to 10. Scoring is taking the mean of items, so the range is 0-10. Lower scores for the scales indicate better quality of life. It provides two summary scales: symptoms and interference. The MDASI takes less than 5 minutes to complete.
Time Frame: Baseline, Day 100, Day 180, 1 year, 2 years
Population: The analyses of the endpoint use the transplanted populations.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CD34 Selected Graft | Post-Transplant Cyclophosphamide | Tacrolimus/Methotrexate Control
Number analyzed (Participants) | 104 | 109 | 114
score on a scale
  Symptoms Score at Baseline: number analyzed (Participants) | 91 | 94 | 98
  Symptoms Score at Baseline | 2 (0.2) | 2 (0.2) | 2 (0.2)
  Symptoms Score at Day 100: number analyzed (Participants) | 79 | 85 | 83
  Symptoms Score at Day 100 | 2 (0.2) | 2 (0.1) | 2 (0.2)
  Symptoms Score at Day 180: number analyzed (Participants) | 71 | 79 | 87
  Symptoms Score at Day 180 | 2 (0.2) | 2 (0.2) | 2 (0.2)
  Symptoms Score at 1 Year: number analyzed (Participants) | 61 | 70 | 80
  Symptoms Score at 1 Year | 2 (0.2) | 1 (0.2) | 2 (0.2)
  Symptoms Score at 2 Years: number analyzed (Participants) | 45 | 53 | 57
  Symptoms Score at 2 Years | 1 (0.2) | 2 (0.2) | 2 (0.2)
  Interference Score at Baseline: number analyzed (Participants) | 90 | 93 | 97
  Interference Score at Baseline | 2 (0.2) | 2 (0.2) | 3 (0.2)
  Interference Score at Day 100: number analyzed (Participants) | 79 | 85 | 81
  Interference Score at Day 100 | 2 (0.2) | 2 (0.2) | 2 (0.2)
  Interference Score at Day 180: number analyzed (Participants) | 71 | 79 | 87
  Interference Score at Day 180 | 2 (0.3) | 2 (0.3) | 2 (0.2)
  Interference Score at 1 Year: number analyzed (Participants) | 61 | 69 | 80
  Interference Score at 1 Year | 2 (0.3) | 2 (0.3) | 2 (0.3)
  Interference Score at 2 Years: number analyzed (Participants) | 45 | 53 | 57
  Interference Score at 2 Years | 1 (0.3) | 2 (0.3) | 2 (0.3)

21. Secondary Outcome: Health-Related Quality of Life (HQL) - PedsQL
Description: HQL will be measured post-transplant using patient-reported survey PedsQL. The PedsQL™ Stem Cell Transplant Module is a 46-item instrument that measures health-related quality of life in children and adolescents undergoing hematopoietic stem cell transplant and is developmentally appropriate for self-report in ages 8 through 18 years. The score ranges from 0 to 100 with higher scores associated with positive outcome.
Time Frame: Baseline, Day 100, Day 180, 1 year, 2 years
Population: The analyses of the endpoint use the transplanted populations.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CD34 Selected Graft | Post-Transplant Cyclophosphamide | Tacrolimus/Methotrexate Control
Number analyzed (Participants) | 0 | 0 | 2
score on a scale
  Pediatric Quality of Life Score at Baseline |  |  | 80.18 (14.94)
  Pediatric Quality of Life Score at Day 100 |  |  | 69.82 (2.75)
  Pediatric Quality of Life Score at Day 180 |  |  | 72.56 (3.05)
  Pediatric Quality of Life Score at 1 Year |  |  | 78.05 (4.27)
  Pediatric Quality of Life Score at 2 Years |  |  | 53.66 (21.34)

ADVERSE EVENTS:
Time Frame: Adverse event reporting and monitoring were conducted throughout the study, up to 2 years.
Description: Adverse event (AE) reporting was conducted according to the BMT CTN's manual of operating procedures (MOP). Unexpected, grade 3-5 AE were reported through an expedited AE reporting system. Expected AEs were reported using National Cancer Institute (NCI)'s Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 at regular intervals and reported in the secondary outcome "Toxicities". All fatal (Grade 5) expected adverse events were reported in an expedited manner.
Arm/Group | CD34 Selected Graft | Post-Transplant Cyclophosphamide | Tacrolimus/Methotrexate Control
All-Cause Mortality (participants affected / at risk) | 42/114 | 27/114 | 30/118
Serious Adverse Events (participants affected / at risk) | 9/114 | 7/114 | 7/118
Other Adverse Events (participants affected / at risk) | 3/114 | 1/114 | 2/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CD34 Selected Graft (N=114) | Post-Transplant Cyclophosphamide (N=114) | Tacrolimus/Methotrexate Control (N=118)
NON CARDIAC CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 1 (1)
NEW MALIGNANCY-RECTAL ADENOCARCINOM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
SEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
SUDDEN CARDIAC ARREST (General disorders) | 1 (1) | 0 (0) | 0 (0)
HOSPITAL ADMISSION FOR INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
DELIRIUM (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
SUDDEN CARDIAC DEATH (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
DEATH (General disorders) | 0 (0) | 1 (1) | 0 (0)
SUPERIOR VENA CAVA SYNDROME (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
EDEMA (General disorders) | 0 (0) | 0 (0) | 1 (1)
COLONIC PERFORATION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
CHOLECYSTITIS (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
FETAL DEATH (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
DISSEMINATED ADENOVIRUS INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
RETROPERITONEAL BLEED (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
GRADE 3 UNEXPECTED WEIGHT LOSS (Investigations) | 0 (0) | 0 (0) | 1 (1)
WORSENING EYESIGHT DUE TO CATARACT (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CD34 Selected Graft (N=114) | Post-Transplant Cyclophosphamide (N=114) | Tacrolimus/Methotrexate Control (N=118)
FOLLICULAR LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
ELEVATED ENDOTOXIN LEVEL (Product Issues) | 1 (1) | 0 (0) | 0 (0)
PLATELET COUNT DECREASE (Investigations) | 1 (1) | 0 (0) | 0 (0)
ELEVATED FERRITIN (Investigations) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-06-22): https://cdn.clinicaltrials.gov/large-docs/50/NCT02345850/Prot_SAP_ICF_000.pdf